CLINICAL TRIAL: NCT00548574
Title: A Phase III, Randomized, Multi-Centre, Double-blind, Double Dummy, Parallel Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Two Doses of SPD476 (Mesalazine) 2.4g and 4.8g Once Daily, With Reference to ASACOL 0.8g Three Times Daily, in Subjects With Mild to Moderate Ulcerative Colitis
Brief Title: Efficacy and Safety of Two Doses of SPD476 (Mesalazine) 2.4g and 4.8g Once Daily, With Reference to Asacol 0.8g Three Times Daily in Subjects With Acute, Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD476-302
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SPD476 is a polymeric matrix formulation that displays both delayed- and extended-release of mesalazine
  Other Names: LIALDA
Drug: Mesalazine
  Other Names: ASACOL

SUMMARY:
The primary objective of the study was to compare the percentage of subjects in remission after 8 weeks of treatment with SPD476, 2.4 g/day once daily vs placebo and SPD476 4.8 g/day once daily versus placebo

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed or relapsing mild to moderate UC (score of 4-10 (inclusive) on the UC-DAI scale, with a sigmoidoscopy score of => 1 and a PGA <=2) with compatible histology
* females eligible if post--menopausal, surgically sterile or if they had a negative urine pregnancy test at screening and were on adequate contraception

Exclusion Criteria:

* subjects with relapsing UC who were in relapse for > 6 weeks prior to baseline
* subjects who relapsed on maintenace therapy with doses of mesalazine => 2g/day
* subjects who had unsuccessfully treated their current relapse with steroids or a mesalazine dose of > 2g/day
* subjects with Crohn's disease, proctitis, bleeding disorders, active peptic ulcer disease, previous colonic surgery, or those at an immediate risk of toxic megacolon or a stool culture positive for enteric pathogens
* subjects who had used systemic or rectal steroids within the last 4 weeks, immunosuppressants wihtin the last 6 weeks or anti-inflammatory drugs on a repeat basis within 7 days prior to the baseline visit
* subjects with hypersensitivity to salicylates and subjects with moderate/severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2003-12-04 (Actual); Primary Completion 2004-10-20 (Actual); Study Completion 2004-10-20 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in remission (UC-DAI score <=1, with scores of 0 for rectal bleeding and stool frequency and a sigmoidoscopy score reduction of 1 point or more from baseline) | 8 weeks

SECONDARY OUTCOMES:
Clinical improvement as defined by a drop of => 3 points from baseline in the overall UC-DAI score | 8 weeks
Change from baseine in UC-DAI score, symptoms, sigmoidscopy score, and PGA | 8 weeks
Clinical remission defined as subjects who scored 0 for both the total stool frequency and the total rectal bleeding score | 8 weeks
Treatment failure defined as unchanged, worsened missing or imcomplete UC-DAI score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Imelda General Hospital Dept of Gastroenterology, Bonheiden, Belgium

REFERENCES:
- [Result] Kamm MA, Sandborn WJ, Gassull M, Schreiber S, Jackowski L, Butler T, Lyne A, Stephenson D, Palmen M, Joseph RE. Once-daily, high-concentration MMX mesalamine in active ulcerative colitis. Gastroenterology. 2007 Jan;132(1):66-75; quiz 432-3. doi: 10.1053/j.gastro.2006.10.011. Epub 2006 Oct 12. PMID 17241860
- See also: FDA-approved labelling information, US only — http://www.lialda.com/Professional/pdf/pi.pdf
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html